CLINICAL TRIAL: NCT06770530
Title: IMPACT - the Introduction of Mycotic Prophylaxis At Cystectomy Trial. Perioperative Mycotic Prophylaxis to Reduce Postoperative Complications Following Cystectomy - a Double-blinded, Placebo-controlled, Randomized Trial
Brief Title: Introduction of Mycotic Prophylaxis At Cystectomy Trial.
Acronym: IMPACT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mie Ynddal, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-506226-36-00
Record Dates: First submitted 2024-05-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-06

CONDITIONS: Cystectomy
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluconazole (Experimental): Intravenous Fluconazole 400 mg single dose in 200 ml saline solution
  Interventions: Drug: Fluconazole
- Isotonic saline solution (Placebo Comparator): Intravenous saline solution single dose 200 ml
  Interventions: Drug: Isotonic saline solution

INTERVENTIONS:
Drug: Fluconazole — 400 mg inravenous Fluconazole, single dose 200 ml
  Arms: Fluconazole
Drug: Isotonic saline solution — Intravenous saline solution, single dose 200 ml
  Arms: Isotonic saline solution

SUMMARY:
This study aims to introduce a perioperative antifungal prophylaxis for patients undergoing cystectomy: surgically removal of the urinary bladder with construction of a urinary diversion. We wish to investigate the effect of antifungal prophylaxis on complications after the operation.

DETAILED DESCRIPTION:
Cystectomy with construction of a urinary diversion, is a major cancer surgery and one of the most complex surgeries in the urological specialty. After cystectomy, the most commonly performed urinary diversion is an ileal conduit, where a section of the terminal ileum is shunted out and connected to the upper urinary tract and a stoma is created. During this procedure, the abdominal cavity is exposed to bacteria and fungus from the ileum. Besides the perioperative contamination, micro-leakage in relation to the anastomosis is suspected to contribute to a local infectious response that may result in postoperative complications as ileal paralysis. Paralytic ileus is a serious complication that affects many patients after cystectomy, resulting in a prolonged length of stay, low quality of life postoperatively, and increased risk of complications such as aspiration, pneumonia, wound rupture, deep venous thrombosis, undernourishment and infections.

Current guidelines support the use of perioperative antibiotics targeting gram-negative and gram-positive bacteria, typically administered as broad-spectrum medicine such as piperacillin/tazobactam or cephalosporins. Regarding fungal infections, emerging data show that 48% of the patients undergoing RC have candida albicans in samples from the terminal ileum. Also, it is well known that fungal infections are highly prevalent in patients undergoing gastrointestinal surgery where it is associated with a high risk of mortality.

Small retrospective studies suggest that the addition of antifungal medicine to perioperative antibiotics can reduce the risk of bowel- and infectious complications after abdominal surgery.

The compelling theoretical and clinical rationale for addition of antifungal prophylaxis to standard-of-care antibiotic prophylaxis for patients undergoing radical cystectomy provides the basis for initiation of a randomized clinical trial representing the highest level of evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Willingness to participate in the study and the ability to understand and sign an informed consent
* Indication for performing cystectomy
* The urinary diversion is limited to the ileal conduit

Exclusion Criteria:

* Patients with contraindications to Fluconazole. This includes allergies and treatment with non-pausable medication that in combination is contraindicated
* Patients in active treatment for mycotic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 90 days from surgery
  Measured by Clavien Dindo III-V classification score. The Clavien Dindo Classification is used to rank the severity of a surgical complication. It consists of seven grades (I, II, IIIa, IIIb, IVa, IVb, V) with I being any deviation from the normal postoperative course and V being death of a patient.

SECONDARY OUTCOMES:
Days Alive and Out of Hospital (DAOH) | 90 days from surgery
  Number of days alive and out of hospital within 90 days from surgery
Time to gastrointestinal function | Postoperatively within 90 days
  First bowel movement
Nasogastric tube placement | Postoperatively within 90 days
  Number of nasogastric tube placements
Length of stay (LOS) | 90 days from surgery
  Duration (days) of primary hospitalization.
Readmission rate | 90 days after surgery
  Number of readmissions
Quality of life (QoL): EORTC QLQ-C30 | Before operation and 90 days after surgery
  Questionnaire from EORTC: European Organization for Research and Treatment of Cancer. All of the scales and single-item measures range in score from 0 to 100. The questionnaires consists of a global health status (high score represents high quality of life), a functional scale (a high score represents a high/healthy level of functioning) and a symptom scale (a high score represents a high level of symptomatology/problems).
Quality of Life(QOL): EORTC QLQ-BLM30 | Before operation and 90 days after
  Questionnaire from EORTC: European Organization for Research and Treatment of Cancer. All of the scales and single-item measures range in score from 0 to 100. The questionnaires consists of a global health status (high score represents high quality of life), a functional scale (a high score represents a high/healthy level of functioning) and a symptom scale (a high score represents a high level of symptomatology/problems).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Røder, MD, PhD, Professor, Principal Investigator — Urological Research Unit, Department of Urology, Rigshospitalet Blegdamsvej 9, 2100 Copenhagen, Denmark; Ulla N Joensen, MD, PhD, Principal Investigator — Urological Research Unit, Department of Urology, Rigshospitalet Blegdamsvej 9, 2100 Copenhagen, Denmark
Locations (1):
- Department of Urology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Maibom SL, Roder MA, Poulsen AM, Thind PO, Salling ML, Salling LN, Kehlet H, Brasso K, Joensen UN. Morbidity and Days Alive and Out of Hospital Within 90 Days Following Radical Cystectomy for Bladder Cancer. Eur Urol Open Sci. 2021 Apr 19;28:1-8. doi: 10.1016/j.euros.2021.03.010. eCollection 2021 Jun. PMID 34337519
- [Background] Andrijasevic N, Ovcaricek S, Butic I, Navratil M, Mili B. Comparison of the effectiveness of two combinations of antibiotic used for perioperative prophylactic therapy during radical cystectomy: A retrospective cohort study. Can Urol Assoc J. 2022 Nov;16(11):E539-E544. doi: 10.5489/cuaj.7859. PMID 35704932
- [Background] Lightner DJ, Wymer K, Sanchez J, Kavoussi L. Best Practice Statement on Urologic Procedures and Antimicrobial Prophylaxis. J Urol. 2020 Feb;203(2):351-356. doi: 10.1097/JU.0000000000000509. Epub 2019 Aug 23. PMID 31441676
- [Background] Villmones HC, Halland A, Stenstad T, Ulvestad E, Weedon-Fekjaer H, Kommedal O. The cultivable microbiota of the human distal ileum. Clin Microbiol Infect. 2021 Jun;27(6):912.e7-912.e13. doi: 10.1016/j.cmi.2020.08.021. Epub 2020 Aug 21. PMID 32835795
- [Background] Prunty M, Rhodes S, Rivero MJ, Callegari M, Jesse E, Arenas-Gallo C, Brant A, Calaway A, Scherr D, Shoag JE. National Adherence to Guidelines for Antimicrobial Prophylaxis for Patients Undergoing Radical Cystectomy. J Urol. 2023 Feb;209(2):329-336. doi: 10.1097/JU.0000000000003069. Epub 2022 Nov 16. PMID 36383758
- [Background] Mitropoulos D, Artibani W, Graefen M, Remzi M, Roupret M, Truss M; European Association of Urology Guidelines Panel. Reporting and grading of complications after urologic surgical procedures: an ad hoc EAU guidelines panel assessment and recommendations. Eur Urol. 2012 Feb;61(2):341-9. doi: 10.1016/j.eururo.2011.10.033. Epub 2011 Oct 29. PMID 22074761
- [Background] Maibom SL, Roder MA, Aasvang EK, Rohrsted M, Thind PO, Bagi P, Kistorp T, Poulsen AM, Salling LN, Kehlet H, Brasso K, Joensen UN. Open vs robot-assisted radical cystectomy (BORARC): a double-blinded, randomised feasibility study. BJU Int. 2022 Jul;130(1):102-113. doi: 10.1111/bju.15619. Epub 2021 Nov 9. PMID 34657367
- [Background] Mitropoulos D, Artibani W, Biyani CS, Bjerggaard Jensen J, Roupret M, Truss M. Validation of the Clavien-Dindo Grading System in Urology by the European Association of Urology Guidelines Ad Hoc Panel. Eur Urol Focus. 2018 Jul;4(4):608-613. doi: 10.1016/j.euf.2017.02.014. Epub 2017 Mar 7. PMID 28753862
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735